CLINICAL TRIAL: NCT00065949
Title: Magnesium Prevention of Brain Injury in Preterm Infants
Brief Title: Magnesium Sulfate to Prevent Brain Injury in Premature Infants
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HD21453; NICHD-13; NICHD-0523; 5R01HD021453 (NIH)
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-05

CONDITIONS: Brain Injuries; Cerebral Palsy
Keywords: Low birthweight infants; Magnesium supplementation; Intracranial hemorrhage; Cystic periventricular leukomalacia; Mental retardation
MeSH Terms: conditions — Brain Injuries; Cerebral Palsy; Intracranial Hemorrhages; Leukomalacia, Periventricular; Intellectual Disability | interventions — Magnesium Sulfate

INTERVENTIONS:
Drug: magnesium sulfate

SUMMARY:
Premature infants are at risk for acute brain injuries and long-term developmental problems such as cerebral palsy (CP). Research suggests that high levels of magnesium at and around the time of birth may decrease the risk of brain injuries. This study will evaluate the effects of giving magnesium to premature infants.

DETAILED DESCRIPTION:
Premature infants weighing less than 1500 grams (3.3 lbs) represent approximately 1.3% of liveborn infants, yet comprise at least 25% of all children who are subsequently diagnosed with CP. Antepartum exposure to magnesium (Mg) may prevent or ameliorate early brain injury (intracranial hemorrhage and cystic periventricular leukomalacia), as well as long-term adverse neurodevelopmental outcomes (CP and mental retardation) in very low birthweight (VLBW) preterm infants. In preliminary studies, short- and long-term neuroprotection were associated with initial serum Mg levels above 3.0 mEq/L. This study will determine whether early abnormal neurosonographic findings and long-term adverse neurodevelopmental outcomes in VLBW premature infants are influenced by different levels of serum Mg achieved during the first week of life.

Infants will be randomized to either "standard" Mg therapy or "high" Mg therapy. Standard Mg therapy consists of no supplemental Mg for the first 3 days of life followed by intravenous magnesium sulfate (MgSO4) aimed at attaining serum Mg levels in the normal range of 1.2-2.3 mEq/L. High Mg therapy consists of using intravenous MgSO4 to maintain higher (nonharmful) serum Mg levels between 3.5-5.5 mEq/L for the first 3 days of life and between 2.5-3.5 mEq/L for the next 4 days. The high Mg infants will subsequently have their serum Mg levels maintained at 2.4+0.3 mEq/L using oral magnesium gluconate for the remainder of their neonatal hospitalization.

Infants will be evaluated for early brain injury with head ultrasound studies 12 to 24 hours after birth, at 2 to 3 day intervals while ventilator support is required, and at weekly intervals until discharge. The infants will subsequently be assessed in the high-risk follow-up clinic for a minimum of 24 months (corrected for degree of prematurity). At 24 months of age, they will be evaluated by a pediatric neurologist for the presence of cerebral palsy. They will be tested serially for problems in early cognition (mental, language, and perceptual ability), as well as fine and gross motor skills.

ELIGIBILITY:
Inclusion Criteria

* Born at 23 to 32 weeks' gestation
* Weighs 500 to 1500 grams (1.1 to 3.3 lbs)
* Requires mechanical ventilation
* Less than 12 hours of age at time of enrollment

Exclusion Criteria

* Multiple congenital anomalies
* Single congenital anomaly of the central nervous system
* Unlikely to be available for duration of the study

Ages: 0 Years to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1987-08; Study Completion 2003-02

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Wiswell, M.D., Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Caddell JL, Graziani LJ, Wiswell TE, Hsieh HC, Mansmann HC Jr. The possible role of magnesium in protection of premature infants from neurological syndromes and visual impairments and a review of survival of magnesium-exposed premature infants. Magnes Res. 1999 Sep;12(3):201-16. PMID 10488476